CLINICAL TRIAL: NCT01096277
Title: Metabolism-independent Vascular Effects of the Dipetidylpeptidase-4-inhibitor Sitagliptin in Patients With Type 2 Diabetes Mellitus
Brief Title: Vascular Effects of Sitagliptin in Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sajoscha A. Sorrentino, MD, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHH_NPH_SS_1/2010; MHH_NPH_SS_1/2010 (Other: Hannover Medical School)
Record Dates: First submitted 2010-03-26; First posted 2010-03-31 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitagliptin (Active Comparator): 100 mg sitagliptin per day for 2 weeks
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): 1 placebo tablet per day for 2 weeks
  Interventions: Drug: Placebo
- Healthy Control (No Intervention): Healthy control subjects
  Interventions: Other: Control

INTERVENTIONS:
Drug: Sitagliptin — oral tablets 100 mg per day for two weeks
  Arms: Sitagliptin
Drug: Placebo — oral tablet, one per day for two weeks
  Arms: Placebo
Other: Control — no intervention
  Arms: Healthy Control

SUMMARY:
Glucagon-like peptide 1 (GLP-1) is a 30-amino acid gut hormone secreted in a nutrient-dependent manner that stimulates insulin secretion and inhibits glucagon secretion and gastric emptying, thereby reducing postprandial glycemia.1,2 GLP-1 is derived from posttranslational proteolysis of preproglucagon, and its peptide sequence is identical in mouse, rat, and human.2,3 After secretion from enteroendocrine L cells, GLP-1(7-36) amide is rapidly degraded by dipeptidyl peptidase-4 (DPP-4) to its N-terminally truncated metabolite GLP-1(9-36), which does not interact with the known GLP-1 receptor.4,5 The diverse actions of GLP-1 include the proliferation, differentiation, and protection from apoptosis of pancreatic β cells and the induction of satiety. GLP-1 also improves memory and learning, stimulates afferent sensory nerves, and has neuroprotective functions.1,6 Furthermore, GLP-1 receptor agonists have been reported to have cardiac and vascular actions in rodents and humans that include effects on contractility, blood pressure, cardiac output,7-10 and cardioprotection.11-14

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of a therapy with the DPP-4-inhibitor sitagliptin on the prognostic relevant endothelial function and endothelial progenitor cells in patients with type 2 diabetes mellitus.

Primary endpoint: Endothelium-dependent vasodilation before and after treatment of patients with type 2 diabetes mellitus with the DPP-4-inhibitor Sitagliptin and placebo treatment respectively.

Secondary endpoint: effect of sitagliptin on mobilization, NO-production and in vivo regenerative capacity of human endothelial progenitor cells before and after treatment of patients with type 2 diabetes mellitus with the DPP-4-inhibitor sitagliptin and placebo treatment respectively

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus

Exclusion Criteria:

* Allergy to sitagliptin
* Treatment with PPAR-gamma agonist

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial function | Before and after two week treatment
  Effect of sitagliptin on endothelium-dependent vasodilation before and after treatment of patients with type 2 diabetes mellitus with the DPP-4-inhibitor sitagliptin and placebo treatment respectively

SECONDARY OUTCOMES:
Effect on EPCs | Before and after two week treatment
  Effect of sitagliptin on mobilization, NO-production and in vivo regenerative capacity of human endothelial progenitor cells before and after treatment of patients with type 2 diabetes mellitus with the DPP-4-inhibitor sitagliptin and placebo treatment respectively

CONTACTS AND LOCATIONS:
Overall Officials: Sajoscha A. Sorrentino, M.D., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany